CLINICAL TRIAL: NCT00849173
Title: Global Study of Women's Health
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090085; 09-CH-0085
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2012-11-26

CONDITIONS: Endometriosis; Infertility; Chronic Pelvic Pain; Tubal Ligation
Keywords: Endometriosis; Infertility; Tubal Ligation; Chronic Pelvic Pain; Quality of Life
MeSH Terms: conditions — Endometriosis; Infertility

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Endometriosis, a condition in which the lining of the uterus grows on nearby tissues, is a common condition that affects women of reproductive age worldwide. The diagnosis of endometriosis is usually made at surgery. The most common symptom is pelvic pain. This pain may occur at the same time as menstrual bleeding, at other times of the cycle, or during or after sexual intercourse. Previous studies reveal the diagnosis of endometriosis is often delayed between 8 and 12 years after the first symptoms. Women with chronic pelvic pain report a lower quality of life. No studies, however, have been conducted to assess whether women with endometriosis-related pelvic pain are affected differently than those with pelvic pain from other or no identifiable causes.

This large-scale study is designed to gather prospective epidemiological data on the impact of and risk factors for endometriosis across countries worldwide. A study of this scale and scope has never been performed; it is anticipated that the study will provide novel insights into the effects of the condition and associated symptoms on women s lives across different countries, as well as explore differences in the effects of various potential risk factors.

This is an international study conducted at more than 20 sites worldwide and coordinated by Oxford University in the United Kingdom. At the National Institutes of Health, 250 premenopausal women between 18 and 45 years of age who are having their first diagnostic laparoscopy or laparoscopy for tubal sterilization will participate. None will have had a prior diagnosis of endometriosis through surgery. Women will be informed about the study when their laparoscopy is scheduled.

Procedures

* Patient completion of an online questionnaire before scheduled surgery. The following will be assessed by the questionnaire:
* Quality of life
* General gynecologic and medical history
* Family history
* General information
* Use of health care services
* Risk factors
* Surgeon completion of questionnaire about surgical findings.
* Follow-up: Women who consent will be contacted every 1 2 years.

DETAILED DESCRIPTION:
This large-scale study is designed to gather prospective epidemiological data on the impact of and risk-factors for endometriosis across countries world-wide. A study of this scale and scope has never been performed; it is anticipated to provide novel insights into the effects of the condition and associated symptoms on women s lives across different countries, as well as explore (differences in) the effects of various potential risk-factors.

Study Design: This is a clinic-based patient survey of prospectively recruited women undergoing a laparoscopy for symptoms suggestive of endometriosis or for tubal sterilization. Descriptive, as well as nested case-control studies will be conducted using information collected from patients in the registry to investigate the impact of endometriosis and associated symptoms, and test etiological hypotheses.

Primary Outcome: The primary purpose of this survey is to collect systematic, comprehensive epidemiological information on the impact of endometriosis among women world-wide, in terms of prevalence, diagnostic delay, quality of life, economic effect indicators, health care utilization, and risk-factors.

Secondary Outcomes: A secondary purpose of the register is to provide a frame-work for future follow-up studies of women diagnosed with endometriosis, allowing the investigation of indicators of effectiveness of different treatment options; long-term quality of life issues, as well as personal and economic (productivity) costs of endometriosis. The multi-center nature of the study should allow variability of endometriosis illness outcomes and associations to be assessed across participating countries.

Statistical Methods:

Basic descriptive analyses will include prevalence estimates according to different age and demographic characteristics, across countries. The analyses of most outcomes will be conducted by comparing women with endometriosis (cases) to those without (controls), both of which will have been recruited through the same process. To avoid bias, cases will be matched to controls on characteristics such as age, country of residence and clinic attended. The analysis of the data will take into consideration this matching; in addition, adjustment for symptoms for which the laparoscopy was indicated (pelvic pain, infertility) will be included. Continuous variables and categorical variables will be analyzed with the appropriate statistical tests.

Duration of Patient Participation: Women are informed about the study at the consultation during which their laparoscopy is scheduled. If they accept to participate, they are asked to fill in an online questionnaire any time before their scheduled surgery. Unless they consent to being contacted sometime in the future for follow-up surveys, their active participation in the study ends. If they wish to participate in future surveys, they will be contacted at most every 1-2 years.

ELIGIBILITY:
* INCLUSION CRITERIA:

A patient who meets all of the following criteria is eligible for the study:

1. Premenopausal female 18 to 45 years of age
2. Attending for her first diagnostic laparoscopy or for laparoscopy for tubal sterilisation
3. Has no previous history of endometriosis diagnosis through surgery

EXCLUSION CRITERIA:

A patient who meets any of the following criteria is ineligible for the study:

1. Already has a surgically-confirmed diagnosis of endometriosis
2. Aged less than18 or greater than 45
3. Aged 18-45 but post-menopausal

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1459 (Actual)
Dates: Start 2009-02-17; Study Completion 2012-11-26

PRIMARY OUTCOMES:
Impact of endometriosis among women worldwide

SECONDARY OUTCOMES:
Provide a frame-work for future studies of women diagnosed with endometriosis which collect long term quality of life issues as well as personal and economic costs of endometriosis.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Stratton, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States